CLINICAL TRIAL: NCT05511922
Title: A Pharmacokinetic Subtrial in Adolescent Patients With Hereditary Angioedema Type I or II Participating in the KVD900-302 Trial
Brief Title: PK Subtrial in Adolescent Patients With HAE Type I or II Participating in the KVD900-302 Trial
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KVD900-302a
Record Dates: First submitted 2022-08-11; First posted 2022-08-23 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hereditary Angioedema
Keywords: KONFIDENT-S; Sebetralstat
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — sebetralstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- KVD900 600 mg (Experimental)
  Interventions: Drug: KVD900 600 mg
- Experimental: KVD900 300 mg (Experimental)
  Interventions: Drug: Drug: KVD900 300 mg

INTERVENTIONS:
Drug: KVD900 600 mg — KVD900 Tablet 600 mg (2 x 300 mg)
  Arms: KVD900 600 mg
Drug: Drug: KVD900 300 mg — KVD900 Tablet 300 mg
  Arms: Experimental: KVD900 300 mg

SUMMARY:
This is a multicenter pharmacokinetic (PK) subtrial to investigate the PK profile of KVD900 (sebetralstat) in adolescent patients 12 to 17 years of age with Hereditary Angioedema (HAE) type I or II.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adolescent patient 12 to 17 years of age at the time of enrollment and during sample collection in this PK subtrial.
* Patient is currently participating in KVD900-302.
* Patient must provide signed informed consent or assent (when applicable), and a legally authorized representative (LAR) must also provide signed informed consent when applicable.
* Patient and LAR are willing and able to provide samples per the requirements of the protocol, including willingness to complete forms and the electronic Diary, obtain and return samples in a timely manner, and obtain samples while within the required age limit.

Exclusion Criteria:

* Patient has a history of any bleeding disorder or currently taking any anti-coagulant or anti-platelet agent.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | Up to 6 hours after IMP administration
Pharmacokinetics - Tmax | Up to 6 hours after IMP administration
Pharmacokinetics - AUC | Up to 6 hours after IMP administration

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — KalVista Pharmaceuticals, Ltd.
Locations (57):
- United States (19):
  - KalVista Investigative Site, Scottsdale, Arizona
  - KalVista Investigative Site, Little Rock, Arkansas
  - KalVista Investigative Site, San Diego, California
  - KalVista Investigative Site, Santa Monica, California
  - KalVista Investigative Site, Centennial, Colorado
  - KalVista Investigative Site, Colorado Springs, Colorado
  - KalVista Investigative Site, Evansville, Indiana
  - KalVista Investigative Site, Overland Park, Kansas
  - KalVista Investigative Site, Louisville, Kentucky
  - KalVista Investigative Site, Chevy Chase, Maryland
  - KalVista Investigative Site, Plymouth, Minnesota
  - KalVista Investigative Site, St Louis, Missouri
  - KalVista Investigative Site, Charlotte, North Carolina
  - KalVista Investigative Site, Cincinnati, Ohio
  - KalVista Investigative Site, Toledo, Ohio
  - Kalvista Investigative Site, Hershey, Pennsylvania
  - KalVista Investigative Site, Dallas, Texas
  - KalVista Investigative Site, Layton, Utah
  - KalVista Investigative Site, Spokane, Washington
- KalVista Investigative Site, Campbelltown, Australia
- KalVista Investigative Site, Vienna, Austria
- KalVista Investigative Site, Sofia, Bulgaria
- KalVista Investigative Site, Montreal, Canada
- France (3):
  - KalVista Investigative Site, Grenoble
  - KalVista Investigative Site, Lille
  - KalVista Investigative Site, Paris
- Germany (4):
  - KalVista Investigative Site, Berlin
  - KalVista Investigative Site, Frankfurt
  - KalVista Investigative Site, Mainz
  - KalVista Investigative Site, Mörfelden-Walldorf
- KalVista Investigative Site, Athens, Greece
- Israel (4):
  - KalVista Investigative Site, Haifa
  - KalVista Investigative Site, Petach Tikvah
  - KalVista Investigative Site, Ramat Gan
  - KalVista Investigative Site, Tel Aviv
- Japan (9):
  - KalVista Investigative Site, Sapporo, Hokkaido
  - KalVista Investigative Site, Chiba
  - KalVista Investigative Site, Hiroshima
  - KalVista Investigative Site, Kawagoe-shi
  - KalVista Investigative Site, Maebashi
  - KalVista Investigative Site, Soka-shi
  - KalVista Investigative Site, Takatsuki-shi
  - KalVista Investigative Site, Tokyo
  - KalVista Investigative Site, Yokohama
- KalVista Investigative Site, Amsterdam, Netherlands
- KalVista Investgative Site, Auckland, New Zealand
- KalVista Investigative Site, Sângeorgiu de Mureş, Romania
- KalVista Investigative Site, Martin, Slovakia
- KalVista Investigative Site, Cape Town, South Africa
- Spain (2):
  - KalVista Investigative Site, Barcelona
  - KalVista Investigative Site, Madrid
- United Kingdom (6):
  - KalVista Investigative Site, Birmingham
  - KalVista Investigative Site, Cambridge
  - KalVista Investigative Site, Cardiff
  - KalVista Investgative Site, Frimley
  - KalVista Investigative Site, Leeds
  - KalVista Investigative Site, London

IPD SHARING:
Plan to Share IPD: No
Data will not be shared until all global regulatory filings are complete.